CLINICAL TRIAL: NCT04012918
Title: Capecitabine in Combination With Aromatase Inhibitor Versus Aromatase Inhibitors, in Hormonal Receptor Positive Recurrent or Metastatic Breast Cancer Patients, Randomized Controlled Study (CONCEPT Trial)
Brief Title: Capecitabine in Combination With Aromatase Inhibitor Versus Aromatase Inhibitors, in Hormonal Receptor Positive Recurrent or Metastatic Breast Cancer Patients, Randomized Controlled Study
Acronym: CONCEPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hesham Elghazaly,MD, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Combined CTH and HT in MBC
Record Dates: First submitted 2019-05-16; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Breast Cancer
Keywords: chemotherapy; aromatase inhibitor; capecitabine; hormonal therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Aromatase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A.I. + Capeciabine (Experimental): Patients will receive Capecitabine 625 mg/m2 bid PO for 14 days to be repeated every 21 days until progression in combination with aromatase inhibitor if postmenopausal, addition of LHRH agonist will be added if premenopausal.
  Interventions: Drug: Capecitabine plus aromatase inhibitor
- A.I (Active Comparator): Patients will receive aromatase inhibitors ( letrozole 2.5 mg PO per day or Anastrozole 1 mg PO per day or aromasin 25 mg PO per day) if post-menopausal, if premenopausal leutnising hormone releasing hormone (LHRH) agonist will be added to the aromatase inhibitor.
  Interventions: Drug: A.I.

INTERVENTIONS:
Drug: Capecitabine plus aromatase inhibitor — Capecitabine 625 mg/m2 bid PO for 14 days to be repeated every 21 days until progression in combination with aromatase inhibitor if postmenopausal, addition of LHRH agonist will be added if premenopausal.
  Arms: A.I. + Capeciabine
Drug: A.I. — aromatase inhibitors ( letrozole 2.5 mg PO per day or Anastrozole 1 mg PO per day or aromasin 25 mg PO per day) if post-menopausal, if premenopausal leutnising hormone releasing hormone (LHRH) agonist will be added to the aromatase inhibitor
  Arms: A.I

SUMMARY:
Women with recurrent or metastatic breast cancer who are hormone receptor positive are candidates for first line hormonal therapy including aromatase inhibitors. In the past few years new combination therapies became available as fulvastrant or palbociclib with letrezole; increasing the progression free survival (PFS). A retrospective study showed that combination of capecitabine with aromatase inhibitors increase PFS as 1st and 2nd line line treatment another prospective study showed the same results. The aim of our study is confirm such data by a randomized controlled trial.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer and the leading cause of cancer death among women worldwide, accounting for 25% of total cancer cases (Globocan, 2012) It ranks as the most prevalent cancer among women in the Middle East and Northern Africa (Ferlay et al., 2015). In Egypt, breast cancer is the most common type of cancer among females (Ibrahim et al., 2014).

Survival of breast cancer patients depends on the disease stage. Most of the patients with localized disease experience long-term disease-free survival. Meanwhile, those who develop metastasis have a 5-year relative survival of only 24% (Siegel et al, 2015). Hormonal receptor positive (HR +ve) represent the most common subset (almost 70%) in both early and advanced disease (Clarke et al., 2012).

It is crucial to determine the menopausal status before initiation of treatment. For HR +ve / Her 2-negative metastatic breast cancer patients who premenopausal; If the patient had Disease free survival (DFS) of 12 months or more, or if she was diagnosed with metastasis de novo, the recommended first line is either ovarian ablation plus tamoxifen or aromatase inhibitor (Cardoso et al., 2017). For postmenopausal patients aromatase inhibitors are recommended with median progression-free survival (PFS) between 8 and 10 months (Bonneterre et al., 2000) and 10 months (Paridaens et al., 2008).

Chemotherapy regimens that are prescribed in hormone receptor-positive patients includes microtubule inhibitors (including taxanes and vinca alkaloids), anthracyclines, gemcitabine, cyclophosphamide and capecitabine. But endocrinal therapy is preferred as long as the patient is not in visceral crisis (Cardoso et al., 2017).

Recently new drugs that increased progression free survival (PFS) has been approved in the treatment of HR +ve metastatic breast cancer (MBC) as fulvastrant (Selective estrogen receptor modulator) (Ellis et al., 2015) and palbocilib (Ck4/6 inhibitor) (Finn et al., 2015) as first line and eveirolimus (mTor inhibitor)(Pritchard et al., 2012) as second line.

The optimum sequence of endocrinal treatment and chemotherapy has not been fully clarified, It is of great importance to bear in mind that the goal of treatment in recurrent and metastatic breast cancer is extending the progression free survival (PFS) and sustaining a good quality of life (Cardoso et al., 2017).

A retrospective study by Shankar et al. that compared between combination of capecitabine and aromatase inhibitor (AI) versus capecitabine alone versus aromatase inhibitor alone showed that the median PFS of first-line treatment was significantly better for the combination with PFS 21 months vs 8.0 months for capecitabine and 15.0 months for AI. For second-line treatment, the PFS was longer in the combination compared with capecitabine and Al groups (18 months vs. 5.0 months vs. 11.0 months, respectively) (Shankar et al., 2015).

Alvarado et al, compared combination aromatase inhibitor plus capecitabine versus capecitabine alone versus aromatase inhibitor alone. The median PFS of first-line treatment was significantly better for the combination (PFS not-reached for combination vs.3.0 m for capecitabine and 13.0 m for AI, p<0.0001). For second-line treatment, the PFS was longer in the combination compared to capecitabine and AI (PFS not reached vs. 6.0 m vs.13.0 m, respectively, p=0-041) (Alvarado et al., 2012).

In China a Phase II trial assessed the use of of metronomic oral capecitabine therapy combined with aromatase inhibitors in postmenopausal metastatic and recurrent breast cancer resistant to first-line aromataseinhibitors and the results showed overall Response Rate (ORR) 70.5% and median PFS 9.57 months (L. Jian-wei et al., 2015). Lee S. Schwartzberg conducted a phase II trial which results showed that fulvastrant with metronomic capecitabine for women with HR-Positive, HER2-Negative MBC has Median PFS was 14.98 months (Schwartzberg et al., 2014).

Capecitabine; being cheaper and more available in economically disadvantaged countries together with the promising results of the previous retrospective trial by Shankar et al and the prospective trial by Alvarado Miranda et al ; further confirmation of such results by a prospective randomized clinical trial is crucial. Currently a phase III trial under the title of "Metronomic Capecitabine Plus Aromatase Inhibitor for First Line Treatment in HR(+), Her2(-) Metastatic Breast Cancer" with the primary results expected to be published on 2021 (Sun Yat-sen University, 2016).

ELIGIBILITY:
Inclusion Criteria:

1. Adult women with locoregionally recurrent or metastatic disease not amenable to curative therapy
2. Eastern Cooperative Oncology Group (ECOG) 0-2
3. Hormone receptor positive
4. No prior systemic anti-cancer therapy for advanced ER+ disease ( hormonal therapy)
5. Measurable disease defined by revised RECIST criteria (version 1.1), or bone-only disease
6. normal laboratory values
7. Postmenopausal or premenopausal with oophorectomy (medical or surgical).

Exclusion Criteria:

1. Patients with advanced, symptomatic, visceral spread that are at risk of life threatening complication in the short term
2. Prior (neo) adjuvant treatment with same aromatase inhibitor type with DFI =< 12 months from completion of treatment.
3. Known uncontrolled or symptomatic central nervous system metastases
4. Second primary malignancy
5. Serious uncontrolled intercurrent infections or intercurrent medical or psychiatric illness
6. unable to swallow tablets, or malabsorption patients.
7. unwilling or unable to comply with study protocol or unable to meet the follow up.
8. patients who researchers considered were not suitable to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — participants are chosen on self-representation of gender identity
Enrollment: 124 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | up to 24 months
  Time from randomization to the first documentation of objective tumor progression or to death due to any cause or Intolerable toxicity.

SECONDARY OUTCOMES:
Adverse events | till progression or up to 24 months whichever earlier
  Detailed Description and grading of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elghazaly, Professor, Principal Investigator — Ain Shams University
Locations (1):
- Clinical oncology department, Faculty of medicine, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Alvarado Miranda, A. et al. (2012) 'Combination treatment with aromatase inhibitor and capecitabine as first- or second-line treatment in metastatic breast cancer.', Journal of Clinical Oncology. American Society of Clinical Oncology, 30(15_suppl), pp. e11016-e11016. doi: 10.1200/jco.2012.30.15_suppl.e11016.
- [Background] Bonneterre J, Thurlimann B, Robertson JF, Krzakowski M, Mauriac L, Koralewski P, Vergote I, Webster A, Steinberg M, von Euler M. Anastrozole versus tamoxifen as first-line therapy for advanced breast cancer in 668 postmenopausal women: results of the Tamoxifen or Arimidex Randomized Group Efficacy and Tolerability study. J Clin Oncol. 2000 Nov 15;18(22):3748-57. doi: 10.1200/JCO.2000.18.22.3748. PMID 11078487
- [Background] Cardoso F, Costa A, Senkus E, Aapro M, Andre F, Barrios CH, Bergh J, Bhattacharyya G, Biganzoli L, Cardoso MJ, Carey L, Corneliussen-James D, Curigliano G, Dieras V, El Saghir N, Eniu A, Fallowfield L, Fenech D, Francis P, Gelmon K, Gennari A, Harbeck N, Hudis C, Kaufman B, Krop I, Mayer M, Meijer H, Mertz S, Ohno S, Pagani O, Papadopoulos E, Peccatori F, Penault-Llorca F, Piccart MJ, Pierga JY, Rugo H, Shockney L, Sledge G, Swain S, Thomssen C, Tutt A, Vorobiof D, Xu B, Norton L, Winer E. 3rd ESO-ESMO International Consensus Guidelines for Advanced Breast Cancer (ABC 3). Ann Oncol. 2017 Jan 1;28(1):16-33. doi: 10.1093/annonc/mdw544. No abstract available. PMID 28177437
- [Background] Clarke CA, Keegan TH, Yang J, Press DJ, Kurian AW, Patel AH, Lacey JV Jr. Age-specific incidence of breast cancer subtypes: understanding the black-white crossover. J Natl Cancer Inst. 2012 Jul 18;104(14):1094-101. doi: 10.1093/jnci/djs264. Epub 2012 Jul 5. PMID 22773826
- [Background] Ellis MJ, Llombart-Cussac A, Feltl D, Dewar JA, Jasiowka M, Hewson N, Rukazenkov Y, Robertson JF. Fulvestrant 500 mg Versus Anastrozole 1 mg for the First-Line Treatment of Advanced Breast Cancer: Overall Survival Analysis From the Phase II FIRST Study. J Clin Oncol. 2015 Nov 10;33(32):3781-7. doi: 10.1200/JCO.2015.61.5831. Epub 2015 Sep 14. PMID 26371134
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] L., J. et al. (2015) 'Phase II clinical trial of metronomic oral capecitabine therapy combined with aromatase inhibitors in postmenopausal metastatic and recurrent breast cancer resistant to first-line aromatase inhibitors', European Journal of Cancer, 51(March), p. S281. doi: 10.1016/S0959-8049(16)30798-5.
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Paridaens RJ, Dirix LY, Beex LV, Nooij M, Cameron DA, Cufer T, Piccart MJ, Bogaerts J, Therasse P. Phase III study comparing exemestane with tamoxifen as first-line hormonal treatment of metastatic breast cancer in postmenopausal women: the European Organisation for Research and Treatment of Cancer Breast Cancer Cooperative Group. J Clin Oncol. 2008 Oct 20;26(30):4883-90. doi: 10.1200/JCO.2007.14.4659. Epub 2008 Sep 15. PMID 18794551
- [Background] Schwartzberg LS, Wang G, Somer BG, Blakely LJ, Wheeler BM, Walker MS, Stepanski EJ, Houts AC. Phase II trial of fulvestrant with metronomic capecitabine for postmenopausal women with hormone receptor-positive, HER2-negative metastatic breast cancer. Clin Breast Cancer. 2014 Feb;14(1):13-9. doi: 10.1016/j.clbc.2013.09.003. Epub 2013 Sep 27. PMID 24268206
- [Background] Shankar A, Roy S, Rath GK, Julka PK, Kamal VK, Malik A, Patil J, Jeyaraj PA, Mahajan MK. Aromatase Inhibition and Capecitabine Combination as 1st or 2nd Line Treatment for Metastatic Breast Cancer - a Retrospective Analysis. Asian Pac J Cancer Prev. 2015;16(15):6359-64. doi: 10.7314/apjcp.2015.16.15.6359. PMID 26434843
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- See also: Sun Yat-sen University (2016) Metronomic Capecitabine Plus Aromatase Inhibitor for First Line Treatment in HR(+), Her2(-) Metastatic Breast Cancer - Full Text View - ClinicalTrials.gov — http://clinicaltrials.gov/ct2/show/NCT02767661
- See also: Globocan (2012) — http://globocan.iarc.fr/Pages/fact_sheets_population.aspx